CLINICAL TRIAL: NCT03039777
Title: Procalcitonin Level as a Surrogate for Catheter-related Blood Stream Bacteremia Among Hemodialysis Patients
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Collaborators: New Jeddah Clinic Hospital (Industry)
Responsible Party: Principal Investigator, Mahmoud Hamada imam, Dr., Benha University
Other Study IDs: 17a1b
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Hemodialysis Catheter Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemodialysis patients frequently develop catheter-related blood stream bacteremia (CRBSI). Procalcitonin is a marker of sepsis in bacterial infection. this study for detection of its role as a surrogacy marker in CRBSI.

DETAILED DESCRIPTION:
Catheter-related blood stream bacteremia is common among hemodialysis patients. Clinically, fever and/or rigors with laboratory indicator of inflammation as leucocytosis and elevated c-reactive protein level are considered as markers for CRBSI before blood culture results became available.

Procalcitonin is a valid indicator of sepsis. In this study, Procalcitonin level will be measured in any patient with suspected CRBSI and correlation will be tested for proved CRBSI by blood cultures.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients with a dialysis catheter
* signs suggestive of CRBSI: fever/chills or leucocytosis with no other site of infection.
* Informed consent signed to be enrolled in the study

Exclusion Criteria:

* Patient with identified cause of fever other than CRBSI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients with clinical signs of CRBSI
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Procalcitonin Level | 2 minutes after start of fever/chills or other symptoms suggesting CRBSI
  Level of serum procalcitonin

OTHER OUTCOMES:
Blood culture (central and peripheral) results | 5 minutes after start of fever/chills or other symptoms suggesting CRBSI
  Blood cultures organism growth results (positive/negative) confirming CRBSI
C Reactive Protein | 2 minutes after start of fever/chills or other symptoms suggesting CRBSI
  Level of C reactive protein
erythrocyte sedimentation rate | 2 minutes after start of fever/chills or other symptoms suggesting CRBSI
  erythrocyte sedimentation rate
Urea Reduction Rate | up to 30 days prior to start of fever/chills or other symptoms suggesting CRBSI
  Urea Reduction rate
creatinine | up to 30 days prior to start of fever/chills or other symptoms suggesting CRBSI
  predialysis Serum creatinine
ferritin | up to 30 days prior to start of fever/chills or other symptoms suggesting CRBSI
  predialysis Serum ferritin
Hemoglobin | up to 30 days prior to start of fever/chills or other symptoms suggesting CRBSI
  Hemoglobin
potassium | up to 30 days prior to start of fever/chills or other symptoms suggesting CRBSI
  predialysis serum potassium
Sodium | up to 30 days prior to start of fever/chills or other symptoms suggesting CRBSI
  predialysis serum sodium

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud H Imam, MD, Principal Investigator — Benha University
Locations (1):
- New jeddah clinic Hospital, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No